CLINICAL TRIAL: NCT04199156
Title: Evaluation of the Non-invasive Blood Pressure Measured at the Ankle During Cesarean Delivery Compared to the Arm: a Prospective Observational Study
Brief Title: Evaluation of Non-invasive Blood Pressure Measured at the Ankle During Cesarean Delivery Compared to the Arm
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Other Study IDs: MS-269-2019
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Non-invasive Blood Pressure; Cesarean Delivery; Spinal Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal anesthesia-induced maternal hypotension during cesarean delivery is hazardous to the mother and the fetus. Prevention of the unfavorable outcomes of maternal hypotension includes various fluid and vasopressor protocols, and requires careful, frequent monitoring of blood pressure during the first 30 minutes after spinal block. Many clinicians set the blood pressure measurement intervals at 1- minute or 2-minutes intervals during the early period after spinal block. it had been reported that hypotension of duration less than 2 minutes is not harmful to the neonate; thus, the minimum inter-measurement intervals for blood pressure readings should be 2 minutes. This high frequency of blood pressure measurements commonly leads to patient dis-satisfaction due to pain as well as impairment of the interaction with the fetus after delivery. Moreover, the blood pressure measurement in the upper limbs could be affected by movement and shivering.

Using the ankle for measurement of non-invasive blood pressure (NIBP) was previously evaluated in normal subjects, and was reported to be feasible; however, its normal range differed from the arm NIBP. Under spinal anesthesia, the lower limb of the mother is neither mobile, nor sensate. Thus, it was previously hypothesized that measurement of blood pressure at the ankle of the mother could improve patient comfort. Darke and Hill had evaluated the accuracy of non-invasive blood pressure at the arm and the ankle during cesarean delivery. Darke and Hill had reported that the degree of bias between the two sites is not acceptable; however, their study did not evaluate the accuracy of ankle NIBP as a trend monitor to trace the changes in maternal blood pressure. The aim of this work is to evaluate the accuracy and precision of ankle NIBP as a trend monitor in mothers undergoing cesarean delivery under spinal anesthesia.

DETAILED DESCRIPTION:
In the preparation room, the parturient will relax in supine position with left uterine displacement by placing a wedge below the right hip. Appropriate size non-invasive blood pressure (NIBP) cuff for the arm and ankle will be chosen according to arm circumference just proximal to antecubital fossa and ankle circumference just above the malleoli, respectively. The cuff's bladder will be directed anteriorly in the arm and in posteriorly in the leg. Simultaneous NIBP measurement of both arms then both ankles will be done. The arm and the ankle with the higher reading will be used for intraoperative NIBP assessment. The baseline reading of the arm and ankle will be obtained as average of 3 reading 2 minutes apart. Simultaneous arm and ankle NIBP measurement will be every 2 minutes from injection of local anesthetic into subarachnoid space till 5 minutes after delivery, then every 5 minutes till the end of surgery. Left uterine displacement will be continued intraoperatively till the delivery. All NIBP measurements will be collected by a research assistant who have no role in parturient management.

Position of the parturient during the spinal anesthesia, drug dosage, fluid management and vasopressor administration will be according to local protocols and the discretion of the attending anesthetist. Intraoperative blood pressure management will be according to the arm NIBP readings

ELIGIBILITY:
Inclusion Criteria:

* full term singleton pregnant women (18-35 years) scheduled for elective cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* Patients with coarctation of aorta,
* cardiac arrythmia,
* impaired cardiac contractility (ejection fraction< 50%),
* congenital heart disease,
* moderate to severe valvular heart disease,
* uncontrolled hypertension,
* known peripheral vascular disease,
* peripartum bleeding,
* body mass index > 35
* Condition which preclude placement of blood pressure cuff on either limb (lymphedema, high risk of developing lymphedema, local skin damage, known vascular stenotic lesion, deep venous thrombosis)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: full term singleton pregnant women (18-35 years) scheduled for elective cesarean delivery under spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
mean bias and agreement between ankle non-invasive blood pressure and arm non-invasive blood pressure | intraoperative (every 2 minutes from injection of local anesthetic into subarachnoid space till 5 minutes after delivery, then every 5 minutes till the end of surgery)
  mmHg

SECONDARY OUTCOMES:
The accuracy of ankle systolic blood pressure to diagnose arm absolute systolic hypotension | intraoperative (every 2 minutes from injection of local anesthetic into subarachnoid space till 5 minutes after delivery, then every 5 minutes till the end of surgery)
  SBP <90 mmHg and < 100 mmHg
The accuracy of ankle systolic blood pressure to diagnose arm relative systolic hypotension | intraoperative (every 2 minutes from injection of local anesthetic into subarachnoid space till 5 minutes after delivery, then every 5 minutes till the end of surgery)
  20% reduction in arm systolic blood pressure
parturient comfort toward arm cuff and ankle cuff | 5 minutes after the surgery
  0= painful, 1=discomfort, 2= comfortable
arm circumference | 5 minutes before the surgery
  cm
ankle circumference | 5 minutes before the surgery
  cm

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Refaat S, Mostafa M, Hasanin A, Rujubali N, Fouad R, Hassabelnaby Y. Accuracy of noninvasive blood pressure measured at the ankle during cesarean delivery under spinal anesthesia. J Clin Monit Comput. 2021 Oct;35(5):1211-1218. doi: 10.1007/s10877-020-00583-y. Epub 2020 Aug 29. PMID 32860553